CLINICAL TRIAL: NCT02514694
Title: LEO 32731 - A Phase I, Single-Blind, Placebo-Controlled, Single and Multiple Oral Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects
Brief Title: LEO 32731 - A Phase I Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LP0058-1114
Record Dates: First submitted 2015-07-08; First posted 2015-08-04 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- LEO 32731 (Active Comparator): Active
  Interventions: Drug: LEO32731
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: LEO32731
  Arms: LEO 32731
Other: Placebo
  Arms: Placebo

SUMMARY:
LEO 32731 ("Study Drug") is an investigational drug which is being developed by LEO Pharma A/S ("the Sponsor") for treatment of psoriasis. The aim (s) of this Study are to determine:

* The safety and tolerability of the Study Drug and any side effects that might be associated with it
* The Study will also measure how much of the Study Drug that gets into the blood and how long time it takes for the body to remove it.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects will, prior to any study related activities, have given their written informed consent to participate in the study and to abide by the study restrictions.
* 2. Subjects will be males or females of non-childbearing potential between 18 and 55 years of age.
* 3. Subjects will have a body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
* 4. For Group C, subjects will be women of non-childbearing potential.
* 5. Subjects must be in good health.

Exclusion Criteria:

* 1. Male subjects who are not willing, or whose partners are not willing, to use appropriate contraception.
* 2. Subjects who have received any prescribed systemic or topical medication within 14 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* 3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* 4. Subjects who have received any medications, including St John's Wort (or other dietary restriction, Section 6.2.3), known to chronically alter drug absorption or elimination processes within 30 days of the first dose administration unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise safety.
* 5. Subjects with a significant history of drug allergy as determined by the Investigator.
* 6. Subjects who have any clinically significant allergic disease (excluding non-active hayfever) as determined by the Investigator.
* 7. Subjects who have a supine blood pressure and supine pulse rate at screening higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 50 bpm, respectively.
* 8. Subjects with a positive urine drug screen or alcohol breath test result at screening or first admission.
* 9. Subjects with, or with a history of, any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological, dermatological or other major disorders as determined by the Investigator.
* 10. Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
* 11. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for HIV antibodies.
* 12. Active tuberculosis or history of incompletely treated tuberculosis, based on medical history or medical report.
* 13. Subjects who, in the opinion of their General Practitioner (GP) or the Investigator, should not participate in the study.
* 14. Subjects with one or more positive faecal occult blood test (immunochemical method) out of 2 assessments at the time between screening and Day-1 check-in.
* 15. Subjects with ≥ 3 bowel movements/day.
* 16. Subjects who have previously taken part in or withdrawn from this study.
* 17. Subjects who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety reported as number of Participants with Adverse Events | 16 days

SECONDARY OUTCOMES:
Pharmacokinetics reported as area under the plasma concentration versus time curve (AUC) | 16 days

CONTACTS AND LOCATIONS:
Locations (1):
- Covance CRU, Leeds, United Kingdom